CLINICAL TRIAL: NCT07020013
Title: Evaluation of the Effectiveness of Day Hospital Care for Adolescents With Anxious School Refusal
Acronym: REPECH
Status: Not yet recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-A00523-46
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: School Phobia
Keywords: School phobia; Anxious school refusal
MeSH Terms: conditions — Phobia, School

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to evaluate the benefit of day care in a child psychiatric hospital on the return to school and on the development of child psychiatric disorders associated with Anxious Social Refusal.

DETAILED DESCRIPTION:
This is a prospective, longitudinal, single-center observational cohort study carried out on a population of patients followed in a day hospital for anxious school refusal.

Participating physicians will have the opportunity to recruit their patients over a 12-month period. All enrolled patients will be followed for a minimum of 10 months. The study will be completed as soon as the last enrolled patient has completed a final assessment.

Aside from the baseline visit, each patient will be assessed only once at 10 months. During each patient visit with the investigating physician, the physician will complete an assessment on the electronic CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 to 18 years
* Patients with anxious school refusal, defined by a score ≥ 41 on the SCREEN scale
* Patients receiving day hospital care
* Patients who have been informed and whose parents (or holder(s) of parental authority) have agreed to their participation in the study and have not objected to the use of their health data

Exclusion Criteria:

* Patients with a mental disability or any other reason that may hinder the understanding or strict application of the protocol
* Patients not affiliated with the French social security system
* Patients under guardianship

Ages: 12 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Population of patients followed in day hospital for anxious school refusal
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Anxious school refusal | Month 10
  The primary endpoint is based on the change in the SCREEN scale score between inclusion and the end of the study. A 20% improvement in this score will be considered as evidence of a benefit from day hospital care on anxious school refusal.

SECONDARY OUTCOMES:
Obsessive-compulsive disorder assessment | Month 10
  The Yale-Brown Obsession-Compulsion Scale (CY-BOCS) is a structured interview that provides an assessment of the severity of obsessive-compulsive symptoms unbiased by the presence or absence of a particular type of obsession or compulsion.
Anxiety disorder assessment | Month 10
  The Spence Children's Anxiety Scale (SCAS) is a 44-item self-report questionnaire. Each item is rated on a 4-point Likert scale, from 0 (never) to 3 (always). No time period is specified for the scope of the questions.
  Six of the 44 items are positive items intended to limit the tendency to respond negatively; they are not included in the overall score.
  The overall score, obtained by adding all 38 items, ranges from 0 to 144. The questionnaire identifies six dimensions of anxiety: Panic Attack and Agoraphobia, Separation Anxiety, Fear of Physical Injury, Social Phobia, OCD, and Generalized Anxiety Disorder.
depressive disorder assessment | Month 10
  The Children's Depression Rating Scale - Revised (CDRS) is a revised version of a questionnaire originally derived from the Hamilton Rating Scale for Depression. The total score is an index of the intensity of depressive symptomatology in children aged 6 to 12 years. It is a 17-item, self-assessment tool, completed by a clinician based on a non-directive interview with the child, and supplemented or corrected, based on clinical judgment, with additional information from the family or teachers.
Post traumatic Stress disorder assessment | Month 10
  The UCLA Child/Adolescent Posttraumatic Stress Disorder Reaction Index was designed for use with school-aged children and adolescents. The DSM-5 version is a semi-structured interview with a clinician that assesses a child's trauma history and the full range of DSM-5 symptoms and diagnostic criteria for posttraumatic stress disorder. This measure consists of several parts: an assessment of different types of trauma, a DSM-5 posttraumatic stress disorder symptom scale including dissociative symptoms, and an assessment of distress and impairment.
Attention Deficit Hyperactivity disorder assessment | Month 10
  The ADHD Rating Scale is a specific assessment tool for ADHD. Consisting of the 18 clinical symptoms involved in diagnosing the disorder in the DSM-IV, it quantifies the severity of the disorder and assesses the various dimensions of the disorder (hyperactivity, inattention, and impulsivity). In most clinical studies, a score of 28 or higher is required to qualify ADHD as significant.
Schooling method | Month 10
  Current schooling method (or planned in the short term) at month 10

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique des 3 cyprès, La Penne-sur-Huveaune, France

IPD SHARING:
Plan to Share IPD: No